CLINICAL TRIAL: NCT06877637
Title: BILe Duct and LIver Cancer: ON-treatment Surveillance of Tumor Evolution And Response to Systemic Treatment
Brief Title: On-treatment Surveillance of Tumor Evolution and Response to Systemic Treatment in Bile Duct and Liver Cancer
Acronym: BILLIONSTARS
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Karin Jirström, Professor, consultant, Region Skane
Other Study IDs: 2024-07592-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC); Cholangiocarcinoma
Keywords: cholangiocarcinoma; hepatocellular carcinoma; bile duct cancer; liver cell cancer; circulating tumor DNA; targeted therapy; tumor heterogeneity; tumor evolution
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor tissue will be obtained from surgical specimens and biopsies, predominantly from formalin-fixed paraffin embedded (FFPE) tissue, but in some cases, fresh tissue will be obtained at surgery for cryopreservation to enable future preclinical studies.
  Plasma, serum and buffy coat will be isolated from blood samples, following standard fractionation, to enable analyses of circulating tumor DNA (ctDNA), and other biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BILLIONSTARS study is a prospective, single arm observational study inviting patients diagnosed with hepatocellular carcinoma (HCC) or cholangiocarcinoma (CCC) who are to be recommended locoregional intervention by surgery, ablation or transarterial chemoembolization and/or antitumoral medical treatment. The aim is to investigate how tumor- and individual-related factors affect response to treatment. To this end, circulating tumor DNA, immune cells and various proteins will be analyzed in repeated blood samples taken before, during and after completion of systemic treatment. When applicable, analyses will also be performed on tumor tissue from resected tumors and biopsies, and in some cases also from autopsies

DETAILED DESCRIPTION:
The BILLIONSTARS study is a prospective, single arm observational study. Patients at Skåne University Hospital in Malmö/Lund and Central Hospital in Kristianstad diagnosed with hepatocellular carcinoma (HCC) or cholangiocarcinoma (CCC) who are to be recommended locoregional intervention by surgery, ablation or transarterial chemoembolization and/or antitumoral medical treatment will be included. A total enrolment of 150 patients is planned.

Before start of treatment, the patients will receive information about the study by a physician and give their written informed consent. Tumor tissue will be obtained from surgical specimens, predominantly from formalin-fixed paraffin embedded (FFPE) tissue, but in some cases, fresh tissue will be obtained at surgery for cryopreservation to enable future preclinical studies. All blood samples will be taken by a dedicated research nurse in conjunction with the treatment visits. Plasma, serum and buffy coat will be isolated from blood samples, following standard fractionation, to enable analyses of circulating tumor DNA (ctDNA), and other biomarkers. Participants will be asked to fill in quality of life questionnaires (EORTC QLQ-C30 and EORTC-QLQ-HCC18/BIL21) at study start, and after three and six months, respectively.

Treatment regimen will follow national guidelines and will not be affected by participation in the study. Radiological and clinical follow ups will be conducted according to clinical protocols or when deemed necessary by the clinician. Primary endpoint is OS, secondary endpoints are progression free survival and change in quality of life (EORTC QLQ-C30+EORTC-QLQ-HCC18/BIL21).

The study will also include research autopsies. Patients are informed and provide their consent for inclusion in this part of the study when they are in a late palliative phase.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Clinically diagnosed intrahepatic Cholangiocarcinoma (iCCC), perihilar Cholangiocarcinoma (pCCC), distal Cholangiocarcinoma (dCCC), gall bladder carcinoma (GBC) or mixed Hepatocellular carcinoma/Cholangiocarcinoma planned to undergo surgery
* Histologically or cytologically confirmed Cholangiocarcinoma (iCCC, pCCC, dCCC, GBC, mixed HCC/CCC) for patients planned to receive palliative systemic treatment or
* Clinically diagnosed Hepatocellular carcinoma (HCC) planned for surgery, ablation or transarterial chemo-embolization. For patients planned to receive systemic treatment histological or cytological confirmation is required except for patients with LI-RADS 5 lesions.

Exclusion Criteria:

* < 18 years of age
* Severe comorbidities
* Inability to comprehend study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Cholangiocarcinoma or Hepatocellular carcinoma at Skåne University Hospital in Malmö/Lund , Sweden, and at Central Hospital in Kristianstad, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of inclusion until the date of death from any cause, assessed up to 60 months"

SECONDARY OUTCOMES:
Progression free survival | From date of inclusion until the date of first documented progression or death from any cause, whichever comes first, assessed up to 60 months.
Impact on quality of life | To be filled out at baseline, at three and at six months.
  Change in quality of life as measured by the form "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Cancer 30 (QLQ-C30). For questions 1-28 the minimum value is 28 and the maximum value is 112, where a higher value indicates worse symptom impact. For questions 29-30 the minimum value is 2 and the maximum value is 14 where a higher value indicates better health status and quality of life.
Impact on quality of life HCC-specific | To be filled out at baseline, at three and at six months.
  Change in quality of life as measured by the form "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Hepatocellular Carcinoma 18 (QLQ-HCC18). For the18 questions the minimum value is 18 and the maximum value is 72, where a higher value indicates worse symptom impact.
Impact on quality of life BTC-specific | To be filled out at baseline, at three and at six months.
  Change in quality of life as measured by the form "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Biliary Tract Cancer 18 (QLQ-BIL21). For the 21 questions the minimum value is 21 and the maximum value is 84, where a higher value indicates worse symptom impact.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Jirström, PhD, MD, professor, Principal Investigator — Region Skåne
Locations (3):
- Sweden (3):
  - Onkologimottagning Central Hospital in Kristianstad, Kristianstad
  - VE Onkologi Skåne University Hospital, Lund
  - VO kirurgi och gastroenterologi Skåne University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falk P, Olsson Hau S, Jacobsen H, Eberhard J, Williamsson C, Jirstrom K. The bile duct and liver cancer: ON-treatment surveillance of tumor evolution and response to systemic treatment (BILLIONSTARS) study. BMC Cancer. 2025 Jun 11;25(1):1017. doi: 10.1186/s12885-025-14429-w. PMID 40500706